CLINICAL TRIAL: NCT04887701
Title: Clinical Outcomes and Safety of a Non-hormonal Medical Device Versus a Sham Device on the Treatment of Vulvovaginal Atrophy (VVA) in Post-Menopausal Women Who Have Failed, Refused, or Are Contraindicated for Hormone Therapy
Brief Title: Non-hormonal Medical Device for Treatment of Vulvovaginal Atrophy (VVA) in Post-Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madorra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLN-201
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Vulvovaginal Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Non-hormonal device therapy (Experimental): Daily non-hormonal device therapy
  Interventions: Device: Non-hormonal vaginal device therapy
- Sham Therapy (Sham Comparator): Daily non-hormonal sham device therapy
  Interventions: Device: Sham vaginal device therapy

INTERVENTIONS:
Device: Non-hormonal vaginal device therapy — Experimental Active Therapy
  Arms: Non-hormonal device therapy
Device: Sham vaginal device therapy — Sham Comparator
  Arms: Sham Therapy

SUMMARY:
Randomized (1:1), double-blind, sham-controlled, 2-arm parallel study comparing effectiveness and safety of non-hormonal medical device versus sham device to treat VVA in post-menopausal women.

DETAILED DESCRIPTION:
After screening and baseline assessment, participants, ages 21 to 65 years of age, will be randomized and followed for a 12-week intervention period. After the primary endpoint evaluation at week 12, each participant in both arms will immediately commence an open label period using an Active device for week 13 to 1 year to collect further effectiveness and safety data.

ELIGIBILITY:
Inclusion Criteria:

* Women with menopause defined by last menstrual period at least 12 months prior to screening, or 6 months of amenorrhea with serum FSH levels > 40 mIU/ml, or 8 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* Sexually active women.
* Participant experiencing subjective moderate-to-severe vaginal pain with sexual intercourse.
* Participant experiencing subjective moderate-to-severe vaginal dryness.
* Gynecological exam confirming vaginal atrophy.
* Willingness to give voluntary written informed consent to participate in the study and comply with protocol requirements.

Exclusion Criteria:

* Use of systemic or local estrogen therapy, currently or in the last 6 months or planned use during the study.
* Use of any other treatment for vaginal atrophy, 6 weeks prior to enrollment or planned during the study period.
* Investigational drugs and also prescription and nonprescription medications/remedies known to treat VVA within 60 days of enrollment or during the study.
* Vaginal stenosis.
* Pelvic floor disorders.
* Prior pelvic radiation therapy including radiation or surgery to the vulva/vagina.
* Active urinary tract, yeast, or other active gynecologic infections.
* Active connective tissue disorders such as lupus or Sjogren's syndrome.
* Active malignancies.
* Diagnosis of vulvodynia or other pelvic pain in the vagina or vulvar area.
* Vulvar dermatoses.
* Laser or radio frequency vaginal rejuvenation treatment or planned treatment during the study.
* Any medical condition that, in the investigator's opinion, would interfere with their participation and/or completion in the study.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 25 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Clinician Assessed Changes in VVA | Baseline to 12 weeks
  Will determine by comparing the mean change between the two arms of the study in clinician assessed changes of VVA by the Vaginal Health Index (VHI). The VHI gives a numerical score (1-5) for each of the 5 parameters measured:
  issue elasticity, vaginal fluid, PH, mucosa, and vaginal moisture.
Patient Reported VAS Score | Baseline to 12 weeks
  Mean change in the Vaginal Assessment Scale (VAS). The VAS is a scale from 0 to 3 with 0 being no symptoms and 3 being severe symptoms.

SECONDARY OUTCOMES:
Responder Rate PGI-I | 12 weeks
  The proportion of patients in the two arms of the study achieving improvement in the patient global impression of improvement (PGI-I), (much or very much improved) at 12 weeks post-treatment.

OTHER OUTCOMES:
Incidence of Adverse Events | 1 year
  Adverse event grading will be done according to the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE)
Patient Satisfaction with Treatment: Likert Scale | 6 months and 1 year
  Patient satisfaction assessed on Likert Scale - a scoring from 0 to 3 (0=not satisfied, 1=neutral, 2=satisfied, 3=extremely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Baber, MD, Principal Investigator — North Shore Private Hospital
Locations (3):
- Australia (3):
  - North Shore Private Hospital, Sydney, New South Wales
  - Goldfields Urology, Bendigo, Victoria
  - Royal Women's Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hickey M, Baber R, Eden J, Brennan J, Bateson D, Goldman M, Rockweiler H, Dreon D. Safety and effectiveness of a novel home-use therapeutic ultrasound device for the treatment of vaginal dryness in postmenopausal women: a pilot study. Menopause. 2023 Apr 1;30(4):383-392. doi: 10.1097/GME.0000000000002157. Epub 2023 Feb 8. PMID 36749915